CLINICAL TRIAL: NCT02654717
Title: Eight Week Study of Treatment With DFD-07 for Actinic Keratosis of the Face and Scalp
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Promius Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFD-07-CD-001
Record Dates: First submitted 2015-12-24; First posted 2016-01-13 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFD-07 cream (Experimental): DFD-07 cream applied twice daily
  Interventions: Drug: DFD-07 Cream
- Placebo cream (Placebo Comparator): Placebo cream applied twice daily
  Interventions: Drug: Placebo Cream

INTERVENTIONS:
Drug: DFD-07 Cream
  Arms: DFD-07 cream
Drug: Placebo Cream
  Arms: Placebo cream

SUMMARY:
The purpose of this study is to see how well DFD-07 works in treating actinic keratosis on the face and scalp during 8 weeks of treatment. The study will also look at any unwanted effects of the study drug.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, the patients have to fulfil all of the following criteria at Visit 1:

1. Written informed consent has been signed and dated prior to any study related procedure or initiation of a wash out period
2. Skin type I, II or III according to Fitzpatrick
3. 5-8 Actinic Keratosis (AK) mild to moderate grade lesions in an approximately 25 cm2 region of scalp, forehead or face that are non-hypertrophic and non-hyperkeratotic
4. 18 years of age or older
5. Female patients of childbearing potential must agree to use contraception during the study which can include abstinence with a secondary contraceptive option should the patient become sexually active. All women of childbearing potential must have a negative urine pregnancy test (test must have a sensitivity of at least 25 IU/ML for human chorionic gonadotropin) at the Baseline Visit. A female is considered of childbearing potential unless she is pre-menarche, postmenopausal with no menses for at least 12 months or surgically sterile. Reliable methods of contraception are hormonal methods or intrauterine devices in use for at least 90 days prior to the Baseline Visit or barrier methods plus spermicide use for at least 14 days prior to the Baseline Visit or a partner who has had a vasectomy at least 3 months prior to the Baseline Visit.
6. ≥ 60 days washout from prohibited medications:

   * Masoprocol
   * 5-Fluorouracil
   * Cyclosporine
   * Retinoids
   * Trichloroacetic Acid/Lactic Acid Peel
   * 50% Glycolic Acid Peel
   * Topical or systemic diclofenac, celecoxib or any other non-sterioda anti-inflammatory drug (however daily low-dose aspirin is allowed, as long as the patient has been on a stable dose, ≤ 100 mg once a day, for 60 days prior to the start of the study.) Note: Patients may use acetaminophen/paracetamol as needed
   * Photodynamic therapy
   * Topical or systemic immunomodulating agents including:

     * Systemic, topical or intralesional interferon
     * Imiquimod (Aldara, Zyclara)
     * Topical ingenol mebutate (Picato)
     * Topical tacrolimus
     * Topical pimecrolimus
     * Sirolimus
     * Cyclosporin
     * Intralesional Bacillus Calmette-Guerin (BCG)
     * Topical coal tar products
     * Topical or systemic corticosteroids

Exclusion Criteria:

Patients who fulfil one or more of the following criteria, will not be eligible for the study:

1. Known or suspected hypersensitivity to any non-steroidal anti-inflammatory drug (NSAID) or a component of the formulation of the study medication
2. Clinical evidence of severe, uncontrolled autoimmune, cardiovascular, gastrointestinal, hematological, hepatic, neurologic, pulmonary or renal disease.
3. Significant history (within the past year) of alcohol or drug abuse
4. Participation in any clinical research study within 60 days of the Baseline Visit.
5. Pregnancy, lactation or plans to become pregnant
6. Concomitant use of cosmetics or other topical drug products on or near the selected treatment area. However, the use of topical sunscreens is allowed.
7. Cosmetic or therapeutic procedures (e.g. laser, peeling, photodynamic therapy) within 2 weeks and within 2 cm of the selected treatment area.
8. Other skin conditions within the selected treatment area (e.g. rosacea, psoriasis, atopic dermatitis, eczema, basal or squamous cell carcinoma or albinism)
9. Use of sun lamps or tanning beds or booths during the 14 days prior to the Baseline Visit or planned use during the study.
10. Any systemic cancer therapy within 6 months of the Baseline Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Site One, Bochum
  - Site Two, Bonn
  - Site Three, Wuppertal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DFD-07 Cream: DFD-07 cream applied twice daily
  DFD-07 Cream
- Placebo Cream: Placebo cream applied twice daily
  Placebo Cream
Period: Overall Study
Arm/Group | DFD-07 Cream | Placebo Cream
Started | 56 | 55
Completed | 50 | 50
Not Completed | 6 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Non-permitted medication | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DFD-07 Cream | Placebo Cream | Total
Number analyzed (Participants) | 56 | 55 | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.0 (9.27) | 72.7 (6.89) | 72.4 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 53 | 49 | 102
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 56 | 55 | 111
Number of Actinic Keratosis lesions [Mean (Standard Deviation); unit: Number of lesions] | 6.1 (1.2) | 6.1 (0.99) | 6.1 (1.09)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Complete Clearance of Lesions
Description: Percent of patients with complete clearance of actinic keratosis (AK) lesions at the end of treatment (8 weeks)
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- DFD-07: Patients treated with DFD07 for 8 weeks
- Vehicle: Pts treated with vehicle for 8 weeks
Arm/Group | DFD-07 | Vehicle
Number analyzed (Participants) | 52 | 51
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline visit until 30 days after the last treatment.
Arm/Group | DFD-07 Cream | Placebo Cream
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/56 | 3/55
Other Adverse Events (participants affected / at risk) | 3/56 | 7/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-07 Cream (N=56) | Placebo Cream (N=55)
Cardiovascular Event (Cardiac disorders) | 0 (0) | 1 (1) — Patient hospitalized with cardiovascular event (no further specification available).
Compression fracture of lumbar vertebral body (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient immobilized with severe lower back pain.
Knee replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Knee replacement for arthritis
B-cell lymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Aggravation of pre-existing B-cell lymphoma
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-07 Cream (N=56) | Placebo Cream (N=55)
Nasopharyngitis (Infections and infestations) | 3 (3) | 7 (7) — Nasopharyngitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No